CLINICAL TRIAL: NCT01858090
Title: Comparison of Intrathecal Levobupivacaine Combined With Sufentanil, Fentanyl, or Placebo for Elective Caesarean Section: A Prospective, Randomized, Double-blind, Controlled Study
Brief Title: Intrathecal Levobupivacaine With Opioids for Caesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nesrin Bozdogan Ozyilkan, Associate Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA08/48
Record Dates: First submitted 2013-05-02; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Elective Caesarean Section Surgeries
Keywords: spinal anesthesia; caesarean section; local anesthetics; levobupivacaine; sufentanil; fentanyl; above 18 years of age; pregnant women; multiparous; nulliparous
MeSH Terms: interventions — Levobupivacaine; Fentanyl; Sufentanil; Ephedrine; Atropine; Propofol; Metoclopramide; Diphenhydramine; Meperidine; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (Placebo Comparator): Control Group, Group C: Spinal anesthesia with levobupivacaine %0.5 (2.2±0.2 ml)+ Serum saline
  Interventions: Drug: Control Group Chirocaine; Drug: Ephedrine; Drug: Atropine sulfate; Drug: Propofol; Drug: Metoclopramide; Drug: Diphenhydramine; Drug: pethidine hydrochloride; Drug: Diclofenac sodium
- Group Fentanyl (Active Comparator): Group Fentanyl, Group F: Spinal anesthesia with levobupivacaine %0.5 (2.2±0.2 ml+fentanyl (10 µg)
  Interventions: Drug: Group Fentanyl; Drug: Ephedrine; Drug: Atropine sulfate; Drug: Propofol; Drug: Metoclopramide; Drug: Diphenhydramine; Drug: pethidine hydrochloride; Drug: Diclofenac sodium
- Group sufentanil (Active Comparator): Group sufentanil, Group S: spinal anesthesia with levobupivacaine %0.5 (2.2±0.2 ml)+ sufentanil (2.5 µg)
  Interventions: Drug: Group sufentanil; Drug: Ephedrine; Drug: Atropine sulfate; Drug: Propofol; Drug: Metoclopramide; Drug: Diphenhydramine; Drug: pethidine hydrochloride; Drug: Diclofenac sodium

INTERVENTIONS:
Drug: Control Group Chirocaine — Control group: Spinal anesthesia with levobupivacaine+Serum Physiologic %0.9 (Total volume 3 mL)
  Other Names: Chirocaine; Chirocaine®, Abbott Laboratories, Ireland; 113/13; 16.12.2002; Serum Physiologic %0.9; Serum Fizyolojik %0.9 10 ml Ampul; Adeka İlac; 8699587751799
  Arms: Control Group
Drug: Group Fentanyl
  Other Names: Fentanyl®, Johnson&Johnson, USA; 110/53; 01.08.2001
  Arms: Group Fentanyl
Drug: Group sufentanil
  Other Names: Sufenta®, Johnson&Johnson, USA; 108/26; 15.08.2000
  Arms: Group sufentanil
Drug: Ephedrine — If systolic blood pressure values decreased more than 20% with respect to the baseline values, or decreased to <100 mmHg, fluid loading and ephedrine (5 mg) were administered.
  Other Names: EFEDRİN HİDROKLORÜR AMPUL 0.05 g, 1 ml; 30.06.1999 - 192/42; OSEL İlaç San. ve Tic. A.Ş. Beykoz/İSTANBUL
Drug: Atropine sulfate — A decrease in heart rate to less than 55 beats/min was considered as bradycardia, and atropine (0.5 mg) was administered
  Other Names: ATROPİN SÜLFAT AMPUL 1/4 mg, 1 ml; 30.06.1999 - 192/9; OSEL İlaç San. ve Tic. A.Ş. Beykoz/İSTANBUL
Drug: Propofol — Intravenous propofol (up to 0.5 mg/kg) was administered if patients had discomfort
  Other Names: Propofol Ampul; Abbott Laboratories, USA; 23.12.1998 - 105/37
Drug: Metoclopramide — Metoclopramide (10 mg IV) was administered for nausea
  Other Names: Metpamid Ampul; Üretici Firma:YENI ILAC VE HAMMADDELERI SANAYI VE TICARET A.S.; Esenyurt/ISTANBUL; 300188-1 BR; Etken Madde(ler):Metoklopramid HCI 10 mg/2 ml
Drug: Diphenhydramine — for severe pruritus
  Other Names: Benison Ampul; Osel İlaç; 8699788750300
Drug: pethidine hydrochloride — pethidine hydrochloride (50 mg IM) was administered as the first analgesic postoperatively
  Other Names: Aldolan ampul; Liba Laboratuarları A.Ş.; 20.12.1985 - 86/29; Gerot Pharmazeutika GmbH, Arnethgasse 3, 1171 Viyana, Avusturya
Drug: Diclofenac sodium — as additional analgesic among cases in which VAS>3(Postoperatively)
  Other Names: Diclomec Ampul 75 mg/ 3 ml; Mecom Saglik Urunleri San. ve Tic. A.S; 8699633759366

SUMMARY:
In this prospective, randomized, double-blind, controlled study, the aim was to compare the effect of adding fentanyl (10 µg) or sufentanil (2.5 µg) to levobupivacaine (2.2±0.2 ml 0.5%) on the intraoperative anesthesia quality, block characteristics, the side effects on the newborn and mother, the duration of postoperative analgesia, and surgeon satisfaction score.

DETAILED DESCRIPTION:
Following the approval of the Baskent University Ethics Committee (KA08/48) and the written informed consents of the patients, 93 pregnant women above 18 years of age without fetal distress/anomaly (gestational pregnancy age ≥ 36 weeks, height ≥ 155 cm, weight ≤110 kg, and fetal weight ≥ 2500 g) and planned American Society of Anesthesiologists (ASA) Physical Status of I to II elective caesarean section surgeries were enrolled. Patients with allergies to any local anesthetic, with a history of hypersensitivity and anaphylactic reactions, who were taken to emergency surgery, and who had preeclampsia were excluded.

Patients were randomized into three groups (Fentanyl Group F, Sufentanil Group S, Control Group C) by a computer, and the demographic data and gestational age of the patients were recorded. No premedications were administered. Following monitoring in all patients (with non-invasive blood pressure, electrocardiogram and pulse oxymeter), Ringer's Lactate solution (15 ml/kg) was administered for 10-15 minutes. Spinal anesthesia was administered with midline approach at the L3-4 interval while the patients assumed a seated position. Spinal blocks were performed by an anesthesiologist blinded to the drug injected, and the drug syringes were prepared immediately before injection by another anesthesiologist who otherwise was not involved in the study. Intraoperative and postoperative assessments were performed by an anesthesiologist blinded to patient allocations and study drugs. 2.2 ml (11 mg) levobupivacaine (Chirocaine®, Abbott Laboratories, Ireland) was administered to patients with heights <163 cm, while 2.4 ml (12 mg) levobupivacaine was administered to patients with heights ≥163 cm (Control Group). 2.2±0.2 ml 0.5% levobupivacaine + 10 µg fentanil (Fentanyl®, Johnson&Johnson, USA) was administered to Group F and 2.2±0.2 ml levobupivacaine + 2.5 µg sufentanil (Sufenta®, Johnson&Johnson, USA) was administered to Group S at rate of 3ml/30 sec. Following intrathecal administration, patients were placed in the supine position, and their heads were slightly elevated. Patients were then brought to a 15-20° left lateral position to prevent aortocaval compression, and oxygen (at 2-4 L/min) was provided with a face mask.

Sensory block was evaluated every two minutes with a pin prick test, while motor block was evaluated with the Bromage scale (0=no motor loss; 1= inability to flex the hip; 2= inability to flex the knee; 3= inability to flex the ankle). Onset times for sensory and motor blocks were recorded. Surgical intervention was initiated when block reached the T5 level. In case sensory block did not attain the T5 level within 20 minutes, general anesthesia was administered.

Duration of sensory block, highest level of sensory block, time to L1-T10 level, time for two-segment and T10 sensory block regression, and the onset and end time of motor block were recorded.

Systolic and diastolic blood pressures (SBP and DBP), heart rate (HR) and oxygen saturations (SpO2) were evaluated every three minutes during the first 15 minutes, and every five minutes afterwards. If systolic blood pressure values decreased more than 20% with respect to the baseline values, or decreased to <100 mmHg, fluid loading and ephedrine (5 mg) were administered. A decrease in heart rate to less than 55 beats/min was considered as bradycardia, and atropine (0.5 mg) was administered. A decrease in the respiratory rate to less than 10/min, and a decrease in oxygen saturation to less than 90%, was considered as indications of respiratory depression. In such cases, support was provided with face mask ventilation.

APGAR scores were evaluated (at minutes 1 and 5) by a pediatrician with no information regarding the groups. For blood gas measurements, samples were obtained from the umbilical cord of newborns.

Intraoperative pain evaluation was performed with the visual analog scale (VAS score; 0= No pain, 10= worst pain possible) while performing surgical incision, uterine incision, and skin closure. In cases where VAS>3, IV fentanyl (50 µg) was administered. Sedation levels were monitored, and propofol (up to 0.5 mg/kg) was administered if patients had discomfort. When patients required more than 50 µg fentanyl and/or 0.5 mg/kg propofol, the block was considered as unsuccessful and general anesthesia was administered. Intraoperative and postoperative nausea, vomiting, pruritus, respiratory depression and other side effects were recorded at the first, second, sixth, and twelfth hours. Metoclopramide (10 mg IV) was administered for nausea, and diphenhydramine (25 mg) was administered for severe pruritus, Surgery procedures were performed by the same surgeon with no knowledge regarding the groups. Surgeon satisfaction score was evaluated according to the sufficiency of muscle relaxation and the provision of adequate surgical conditions (0= pair, 1= fair, 2= good, 3= excellent).

The time of first analgesic requirement was recorded for the patients, and pethidine hydrochloride (50 mg IM) was administered as the first analgesic. Following this, analgesic treatment was continued with diclofenac sodium (75 mg IM) as additional analgesic among cases in which VAS>3. Diclofenac sodium requirement during the first 24 hours were recorded.

Statistical Analysis Sensory block duration was used as main end-point for statistical analysis. Power analysis based on previous studies14,15 indicated that the minimum number of patients required for 80% power (α=0,05, β=0,20) was 24 per group for detecting 25% difference in sensory block duration. Statistical analysis was performed using SPSS version 17.0 (SPSS Inc, Chicago, Illinois). Categorical measurements were recorded as numbers and percentages, continuous measurements with mean and standard deviation (Mean±SD), and also with the median (minimum-maximum) where necessary. In the comparison of categorical variables, the chi-square test or the Fischer's exact test were used. The ANOVA test was used for distributions, in the comparison of continuous measurements between the groups, while the Kruskal-Wallis test was used for parameters without normal distribution. Hemodynamic data were analyzed with repeated measure analyses. Values of p<0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* above 18 years of age
* gestational pregnancy age ≥ 36 weeks
* height ≥ 155 cm
* weight ≤110 kg
* fetal weight ≥ 2500 g)
* American Society of Anesthesiologists (ASA) Physical Status of I to II
* elective caesarean section surgeries were enrolled.

Exclusion Criteria:

* Local anesthetic allergy
* history of hypersensitivity and anaphylactic reactions
* emergency surgery
* preeclampsia

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the effect of adding fentanyl or sufentanil to levobupivacaine (2.2±0.2 ml 0.5%) on intraoperative anesthesia quality block characteristics side effects on newborn and mother,duration of postoperative analgesia,surgeon satisfaction score | during caesarean section and postoperative first 24 hours

OTHER OUTCOMES:
The time of first analgesic requirement | Postoperative first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anis Aribogan, Prof., MD, Study Director — Baskent University School of Medicine
Locations (1):
- Baskent University School of Medicine Adana Teaching and Research Hospital, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Karaman S, Kocabas S, Uyar M, Hayzaran S, Firat V. The effects of sufentanil or morphine added to hyperbaric bupivacaine in spinal anaesthesia for caesarean section. Eur J Anaesthesiol. 2006 Apr;23(4):285-91. doi: 10.1017/S0265021505001869. Epub 2006 Jan 27. PMID 16438758
- [Derived] Bozdogan Ozyilkan N, Kocum A, Sener M, Caliskan E, Tarim E, Ergenoglu P, Aribogan A. Comparison of intrathecal levobupivacaine combined with sufentanil, fentanyl, or placebo for elective caesarean section: a prospective, randomized, double-blind, controlled study. Curr Ther Res Clin Exp. 2013 Dec;75:64-70. doi: 10.1016/j.curtheres.2013.09.003. PMID 24465046